CLINICAL TRIAL: NCT01444690
Title: Dimiracetam in Painful Neuropathies Affecting AIDS Patients. A Double-blind, Placebo-controlled, Parallel-group, Randomised, Multi-centre Study
Brief Title: Dimiracetam in Painful Neuropathies Affecting AIDS Patients
Acronym: DIPANAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neurotune AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NT-004-DIPANAP
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Antiretroviral therapy; Acquired Immunodeficiency Syndrome/complications*; Anti-HIV Agents/adverse effects
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dimiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Dimiracetam 400 mg capsules
  Interventions: Drug: Dimiracetam
- Pseudo-placebo (Placebo Comparator): Dimiracetam 25 mg capsules
  Interventions: Drug: Dimiracetam 25 mg

INTERVENTIONS:
Drug: Dimiracetam — Capsules for oral administration twice daily
  Arms: Active
Drug: Dimiracetam 25 mg — Inactive dose level in capsules administered orally twice daily
  Arms: Pseudo-placebo

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability of orally administered dimiracetam for 10 weeks to AIDS patients under treatment with antiretroviral agents presenting a disease and /or treatment related neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged 18-75 years inclusive;
* females of child-bearing potential only if agreeing prior to screening to use a medically accepted method of contraception, i.e., oral or injectable hormonal contraceptive with a second method of birth control, medically prescribed intrauterine device (IUD), or double barrier method (condom in combination with spermicidal). Females, who are not currently sexually active, only if agreeing and consenting to use one of the above-mentioned methods in case they become sexually active while participating in the study;
* females of not child-bearing potential only if permanently sterilised or if in post-menopausal status, only if they have been in this status for at least 2 years; females of not child-bearing potential are exempted from the requirement for use of contraception;
* HIV-positive patients treated with ARTs;
* CD4+ cell count > 200/μL at the screening;
* patients affected by current neuropathic pain likely to be ART treatment related. The diagnosis shall be made by a physician and based on history, clinical and/or laboratory findings in accordance with the taxonomy of the diagnostic criteria documented in the International Association for the Study of Pain (IASP) Classification of Chronic Pain;
* naïve neuropathic patients or non-responders (residual pain ≥40 mm on the VAS) to standard neuropathy treatments. Drugs for neuropathic pain (NP) must be stopped at screening visit;
* pain intensity ≥40 mm on the VAS at screening;
* pain intensity ≥40 mm on the VAS as the mean of the values collected on the last 4 days prior to the start of treatment (baseline VAS);
* life expectancy of at least 6 months;
* ability to comprehend the full nature and purpose of the study, including possible risks and side effects;
* ability to co-operate with the Investigator or designee and to comply with the requirements of the entire study

Exclusion Criteria:

* pregnant or lactating females;
* presence of active AIDS-defining opportunistic infections (with the exception of tuberculosis) or malignant neoplasia requiring treatment at study entry or Kaposi's sarcoma or another malignant neoplasia likely to require chemotherapy;
* any clinically significant underlying disease, according to the Investigator's clinical judgment;
* history of psychosis (e.g. schizophrenia or psychotic depression) or major depression (requiring treatment);
* any current DSM-IV Axis I diagnosis including dementia, depression, psychosis, anxiety disorders, mental retardation;
* participation in the evaluation of any investigational drug within 3 months prior to screening (6 months if for treatment of neuropathic pain)
* treatment with neurostimulating devices such as spinal cord stimulation (SCS), acupuncture, homeopathic remedies for pain or any kind of surgical treatment or blockade for the pain in the 4 weeks prior to screening;
* treatment with any drug for neuropathic pain (NP) after the screening visit;
* requirement of more than 2 transfusions / month to achieve haemoglobin level > 8 g/dL;
* history of alcohol abuse (no more than 4 drinks in a day and 14 drinks in a week for men or 3 drinks per day and 7 drinks in a week for women as defined according to both NIAAA and USDA dietary guidelines) or drug abuse during the last 3 mo prior to screening;
* Less than 1 VAS assessment per day for each of the last 4 days.
* history of allergic response to neuropathic treatments or history of anaphylaxis or allergic reactions to drugs in general;
* any abnormality that the Investigator deems to be clinically relevant, either on medical history, physical examination, ECG or in diagnostic laboratory test;
* subjects likely to be non-compliant or uncooperative during the study according to the Investigator or designee's judgement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured on 100 mm VAS | 71 days
  Change from baseline in pain intensity as measured on VAS
Pain intensity as measured with Total Symptom Score (TSS) | 71 days
  Change from baseline as measured with TSS

SECONDARY OUTCOMES:
Adverse events | 78 days
  Comparison of AE frequency between treatment groups
Number needed to treat | 71 days
  NNT needed to obtain a >60% pain relief from the initial score recorded on the VAS and TSS at study entry
CD4+ cell count | 78 days
  comparison of CD4+ cell count vs. baseline within and between treatment groups
HIV viral load | 78 days
  comparison of HIV viral load vs. screening within and between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Rugerro Fariello, MD, Study Director — Neurotune AG
Locations (1):
- Neurotune AG, Lugano, Switzerland